CLINICAL TRIAL: NCT03461250
Title: Chronic Hepatitis C in Chronic Hemodialysis Recipients - An Observational Study
Acronym: (CHINCHERO)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asociacion para el Estudio del Higado (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, P. Martin Padilla-Machaca, MD, Asociacion para el Estudio del Higado
Other Study IDs: AsociacionPEH
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: HCV Infection
Keywords: HCV infection; hemodialysis; HCV genotype; Liver Fibrosis stage
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCV serology negative in HD: Risk factors
  Interventions: Diagnostic Test: HCV serology
- HCV serology positive in HD: Risk factors HCV viral load HCV genotype Liver elastography by Fibroscan
  Interventions: Diagnostic Test: HCV serology

INTERVENTIONS:
Diagnostic Test: HCV serology — Apply CRF to identify risk factors for HCV infection. In patients with positive HCV serology measure the level of viral load and HCV genotype by PCR Abbott-real time and determine the stage of liver fibrosis by elastography (Fibroscan)
  Other Names: HCV viral load; HCV genotype; Liver fibrosis stage by Fibroscan

SUMMARY:
This is an observational study of cases of chronic hepatitis C and negative HCV controls in adults receiving chronic hemodialysis at the National Renal Health Center (NRHC) -EsSalud in Lima - Peru.The NRHC provides specialized health care, including hemodialysis, to people with advanced kidney disease from all the districts of Lima.

Study population: By December 2017, there were 293 adults receiving chronic hemodialysis at the NRHC-EsSalud.

All adult patients receiving chronic hemodialysis at the NRHC-EsSalud will be invited to participate.

Primary objective: Characterize HCV disease in patients receiving chronic hemodialysis at the NRHC-EsSalud.

Secondary objective: Identify factors associated with an increased risk of HCV infection.

Inclusion criteria:

Age > 18 years Receive chronic hemodialysis (for at least 6 consecutive months) at the NRHC.

Exclusion criteria:

• Inability to provide informed consent. To comply with the primary objective of the study, samples from volunteers with HCV serology confirmed in Roe Clinic Laboratory (cases) will be subjected to additional tests: HCV viral load followed by determination of the HCV genotype by using the Abbott m2000 real-time PCR system capable of identifying genotypes 1 (1a and 1b), 2, 3, 4 , 5 and 6, using fluorescent probes of oligonucleotides specific for each genotype .

In addition to these lab tests, volunteers will have a Fibroscan test performed at a local provider, with the Fibroscan Model 402 with E and XL probes.

The information will be collected in a Case Report Form (CRF), which will be filled out by study staff. The source of clinical information will be primarily the clinical history of the NRHC - EsSalud. The source of information on the results of the auxiliary tests will be obtained from the results issued by Roe Clinic Laboratory and by the image center of the Delgado Clínic.

Protection of Human Subjects:

The protocol and informed consent will be reviewed and approved by the Ethics Committee of the NRHC. No study procedure will be carried out if the volunteer has not given his or her written consent. All reasonable precautions will be taken to protect the privacy of the volunteer's information, whose data will be identified only through a code. Researchers will keep the study folders in a locked cabinet in a safe place

DETAILED DESCRIPTION:
Epidemiological Data

It is estimated that chronic infection with the chronic hepatitis C virus (HCV) affects approximately 180 million people worldwide (1). It has surpassed HIV infection as the leading cause of death from viral infection in multiple countries including the United States (2). Complications of chronic HCV occur after several years and include cirrhosis, liver failure, need for liver transplantation, and hepatocellular carcinoma. Complications of cirrhosis include portal hypertension, spontaneous bacterial peritonitis, gastrointestinal bleeding, and hepatic encephalopathy, among others (3). There are also multiple extrahepatic manifestations of the disease such as uveitis, cryoglobulinemia, autoimmune thrombocytopenic purpura, membranoproliferative glomerulonephritis, Porphyria Cutaneous Tarda (PCT), among others (4). Consequently, HCV represents a major cause of health care expenses.

In Peru, the prevalence of HCV in the general population is estimated at less than 1%. While people receiving multiple blood transfusions and health workers are known risk groups, the highest prevalence - 59% (5,6) - has been reported in people receiving chronic hemodialysis.

Previously, patients with chronic kidney disease - stage 5 received blood transfusions for the treatment of anemia associated with this disease so it was considered an important risk factor, which has decreased with the use of erythropoietin (EPO). Currently, the most important risk factor in dialysis is nosocomial transmission related to the biosecurity practices used.

New era in the treatment of HCV: The HCV treatment standard in Peru has been pegylated interferon +/- ribavirin, however, its use in patients on hemodialysis has been limited due to its low efficacy and unfavorable safety profile. There is a clear need for new HCV treatments that are effective and well tolerated.

In recent years there has been a significant improvement in drugs and drug combinations for the treatment of HCV. The current treatments are oral interferon-free schedules, which combine 2 or more medications called direct acting agents (DAA). DAAs schemes are highly effective and well tolerated, with cure rates above 90% even in patients who have traditionally been difficult to treat. The metabolism of DAAs varies among the different classes, being that only a few have indication of use in people receiving hemodialysis (7).

Preliminary local data: The Social Security of Peru (EsSalud) is the second largest public health system in the country, which has been treating most people who require chronic hemodialysis in Peru. The National Renal Health Center (NRHC) of the Social Security of Peru (EsSalud) provides specialized health care, including hemodialysis, to people with advanced kidney disease from all the districts of Lima. Currently they serve 293 people on chronic hemodialysis. Because the NRHC routinely performs the serology test for HCV, they have identified 124 patients (42.32% of all patients on hemodialysis at the NRHC) with positive serology for HCV and 12 additional patients (4% of patients in hemodialysis) who have mixed infection with HCV and with the hepatitis B virus (HBV). Those 136 patients with chronic hepatitis C will have already developed or will eventually develop the complications of the disease that will result in a high economic burden for EsSalud.

Since Peru is entering the era of interferon-free HCV treatments, with regimens that are effective and safe in hemodialysis patients, there is the potential to implement interventions that reduce or even eradicate HCV infection from hemodialysis programs.

Significance: The characterization of HCV disease in chronic hemodialysis patients in terms of genotype, viral load, and degree of liver fibrosis will be of key importance to understand the burden of disease and to define priorities and interventions. Additionally, understanding the risk factors associated with chronic HCV infection in this setting will inform decision makers so that they can optimize policies and procedures to keep hemodialysis programs free of this infection.

METHODS:

Study design:

This is an observational study of cases of chronic hepatitis C and negative HCV controls in adults receiving chronic hemodialysis at the NRHC-EsSalud.

Objectives of the study:

* Primary objective: Characterize HCV disease in patients receiving chronic hemodialysis at the NRHC-EsSalud.
* Secondary objective: Identify factors associated with an increased risk of HCV infection.

Inclusion criteria:

* Age > 18 years
* Receive chronic hemodialysis (for at least 6 consecutive months) at the NRHC-EsSalud

Exclusion criteria:

• Inability to provide informed consent

Procedures of the study:

All adult patients receiving chronic hemodialysis at the NRHC-EsSalud will be invited to participate in the study. Before conducting any study procedure, volunteers will sign a consent form approved by the local ethics committee. For volunteers who have signed the informed consent will proceed to make the review of their clinical history will be invited to provide a blood sample for HCV serology to be held in the Roe Clinic Laboratory. Although patients in hemodialysis in the NRHC-EsSalud undergo periodic evaluation with HCV serology, performing the HCV serology in Roe Clinic Laboratory as a procedure of this study will provide a confirmation of the results with a standardized method (an automated test of third-generation electrochemical-luminescence, made with the Cobas® e 601 immunoassay analyzer from Roche Diagnostics).

After determining the serology result for hepatitis C in each patient, proceed according to the following flow diagram:

Chronic hemodialysis in adults: Informed consent

HCV + :

Main objective: Define HCV disease Clinical chart review HCV genotype HCV viral load Fibroscan

HCV -:

Secondary objective: Define HCV risk factors Clinical chart review Electronic data review

To comply with the primary objective of the study, samples from volunteers with HCV serology confirmed in Roe Clinic Laboratory (cases) will be subjected to additional tests: HCV viral load followed by determination of the HCV genotype. The total blood volume to be obtained from each volunteer will not be greater than 16 ml.

The viral load of HCV will be quantified by using the Abbott m2000 real-time Polymerase Chain Reaction (PCR) system. Samples from volunteers with positive serology for HCV and detectable viral load will be analyzed to determine the HCV genotype using the Abbott RealTime HCV Genotype II test, capable of identifying genotypes 1 (1a and 1b), 2, 3, 4 , 5 and 6, using fluorescent probes of oligonucleotides specific for each genotype.

In addition to these lab tests, volunteers will have a Fibroscan test performed at a local provider, with the Fibroscan Model 402 with E and XL (extra large) probes.

To comply with the secondary objective, both cases and controls (volunteers with negative serology for HCV in Roe Clinic Laboratory) will be invited. A predefined format will be applied to collect information on cases and controls including: date of birth, sex, time since the first hemodialysis, date of the first positive local serology, frequency of dialysis, time since the first hemodialysis at the NRHC-EsSalud , number of centers where hemodialysis was attended, history of surgery (yes / no, and type of surgery) before the diagnosis of HCV, history of blood transfusions or by-products (yes / no, and number) before diagnosis of HCV, type of venous access for hemodialysis (AV / catheter fistula), use of dedicated hemodialysis machines (yes / no), use of individual filters (yes / no), comorbidities (such as diabetes mellitus, HIV infection, and other conditions of immunosuppression), history of transplantation, number and type of sexual partners, and history of intravenous drug use.

The study is expected to be completed within six months of its local approval.

Statistical considerations:

Study population: By December 2017, there were 293 adults receiving chronic hemodialysis at the NRHC-EsSalud. Given that the patients of this center are tested for HCV serology every six months, it is known that 124 (42.3%) patients have HCV infection and 12 additional patients have co-infection with HBV and HCV, giving a total of 136 infected with HCV (general prevalence of 46.41%). The remaining 157 patients have negative serology for HCV. These numbers may vary when the serology confirmation results are known (done as a procedure in this study).

All adult patients receiving chronic hemodialysis at the NRHC-EsSalud will be invited to participate, therefore an estimate of sample size does not correspond.

The collected data will be analyzed with Statistical Package for the Social Sciences (SPSS). Descriptive statistics will be applied, including medians and means ± Standard Deviation (SD). Proportions will be used for the categorical variables. Unpaired T-test will be used to compare medians of time in dialysis and age. Poisson regression (bivariate) will be used to evaluate associations of variables with HCV infection. Multivariate Poisson regression analysis will be used to model the associations between the explanatory variables detected as significant in the univariate analysis. The level of statistical significance for the univariate analysis will be 0.10 and for the multivariate it will be 0.05.

Collection and Data Management:

The information will be collected in a Case Report Form (CRF), which will be filled out by study staff. The source of clinical information will be primarily the clinical history of the NRHC-EsSalud. The source of information on the results of the auxiliary tests will be obtained from the results issued by Roe Clinic Laboratory and by the image center of the Delgado Clinic.

Protection of Human Subjects:

The protocol and informed consent will be reviewed and approved by the Ethics Committee at the NRHC. No study procedure will be carried out if the volunteer has not given his or her written consent. All reasonable precautions will be taken to protect the privacy of the volunteer's information, whose data will be identified only through a code. Researchers will keep the study folders in a locked cabinet in a safe place.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years
* Receive chronic hemodialysis (for at least 6 consecutive months) at the NRHC. EsSalud

Exclusion Criteria:

* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on chronic hemodialysis for at least 6 consecutive months at the NRHC. EsSalud. Lima. Peru.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
Characterize HCV disease in patients with chronic hemodialysis at the NRHC-EsSalud | 6 months
  Determine risk factors HCV infection with CRF and clinical charts review, level of viral load and HCV genotype and liver stage fibrosis by Fibroscan.

CONTACTS AND LOCATIONS:
Overall Officials: P.Martin Padilla, MD, Principal Investigator — Asociacion para el Estudio del Higado

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ly KN, Xing J, Klevens RM, Jiles RB, Ward JW, Holmberg SD. The increasing burden of mortality from viral hepatitis in the United States between 1999 and 2007. Ann Intern Med. 2012 Feb 21;156(4):271-8. doi: 10.7326/0003-4819-156-4-201202210-00004. PMID 22351712
- [Background] Marcellin P. Hepatitis C: the clinical spectrum of the disease. J Hepatol. 1999;31 Suppl 1:9-16. doi: 10.1016/s0168-8278(99)80368-7. PMID 10622554
- [Background] Cacoub P, Comarmond C, Domont F, Savey L, Desbois AC, Saadoun D. Extrahepatic manifestations of chronic hepatitis C virus infection. Ther Adv Infect Dis. 2016 Feb;3(1):3-14. doi: 10.1177/2049936115585942. PMID 26862398
- [Background] Sanchez JL, Sjogren MH, Callahan JD, Watts DM, Lucas C, Abdel-Hamid M, Constantine NT, Hyams KC, Hinostroza S, Figueroa-Barrios R, Cuthie JC. Hepatitis C in Peru: risk factors for infection, potential iatrogenic transmission, and genotype distribution. Am J Trop Med Hyg. 2000 Nov-Dec;63(5-6):242-8. PMID 11421371
- [Background] Mendez Chacon P, Vidalon A, Vildosola H. [Risk factors for hepatitis C in hemodialysis and its impact on the waiting list for kidney transplantation]. Rev Gastroenterol Peru. 2005 Jan-Mar;25(1):12-8. Spanish. PMID 15818418
- [Background] Fabrizi F, Messa P. Therapy of hepatitis C by direct-acting anti-virals: the end of HCV in dialysis population? Expert Rev Clin Pharmacol. 2015;8(6):785-93. doi: 10.1586/17512433.2015.1086266. Epub 2015 Sep 12. PMID 26365524
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- See also: HCV epidemiology — http://www.who.int/mediacentre/factsheets/fs164/en/